CLINICAL TRIAL: NCT06785103
Title: Transformative Approaches to Rapidly and Efficiently Test Demand Creation Interventions to Promote HIV Retesting in Adults at Increased Risk of HIV
Brief Title: IBIS Megastudy- Pilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: On 5/1/25, the US NIH issued Notice: NOT-OD-25-104, which prohibited foreign subawards from being nested under a parent grant. Our pilot trial was scheduled for renewal on 8/1/25, and the NOA was delayed. Without funding, we had to halt the trial.
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Pennsylvania (Other); Kenya Medical Research Institute (Other); Infectious Diseases Research Collaboration, Uganda (Other); University of California, Berkeley (Other); Makerere University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23-39197; R01MH132438 (NIH)
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: behavioral economics; "nudge" interventions; Uganda; Kenya; HIV retesting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- HIV Risk Assessment (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Emphasize that a negative test doesn't mean that previous behavior(s) weren't high-risk
  * Enable people to re-assess their own personal risk at a later/future date
  * Suggest risk behaviors to reflect on
  * If participant has engaged in one or more behaviors, emphasize their need to re-test
  Interventions: Behavioral: Risk assessment messaging
- U=U messaging (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  Explain benefits of finding out your HIV-positive status as early after infection as possible and start treatment as soon as possible. These benefits include:
  * Prevent transmission of HIV to anyone
  * Live a normal life, with freedom in sexual choices and ability to start a family
  Interventions: Behavioral: U=U messaging
- Healthy Living (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Illustrate how regular HIV testing is one part of a healthy lifestyle
  * Use examples to connect/compare retesting to other ways to protect/improve overall health
  Interventions: Behavioral: Healthy Living messaging
- Community benefits (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Emphasize that regular testing keeps the participant's community safe and healthy by reducing chances of transmitting HIV unknowingly
  * Call for responsibility- the participant to do their part for the community; they are an integral part of the solution
  Interventions: Behavioral: Community benefits messaging
- Fresh start effect (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Using a specific moment in time (like a resolution, start of a new month, etc.) to motivate a healthy behavior (i.e. a "fresh start" moment)
  * emotional unburdening of resolving uncertainty (not knowing one's status is more stressful than knowing one's status, whether positive or negative, and being able to take healthy steps after knowing if the status is negative or positive)
  Interventions: Behavioral: Fresh start effect
- Education-based #1 (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Provide basic scientific information about HIV virus and transmission
  * Mention private, individual benefits of early HIV treatment
  Interventions: Behavioral: Education-based messaging (#1)
- Education-based #2 (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Increase attention to HIV re-testing reminder through interactive trivia questions
  * Correct or reinforce understanding about HIV prevention, transmission, and retesting
  Interventions: Behavioral: Education-based #2 messaging (gamification)
- Default appointment (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Having a set appointment will reduce uncertainty about availability for retest visit
  * Having an opt-out option for the future retesting appointment
  * A planning prompt to be specific about the participant's future plan for retesting
  * Gentle/soft commitment: by picking a date, mentally agree to come back to retest
  Interventions: Behavioral: Default appointment messaging
- Reserved for you (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Make participant aware that the test is available, and the clinic is welcoming the participant to receive it
  * "VIP status-" the participant is lucky/special to have this opportunity
  Interventions: Behavioral: Reserved for you messaging
- Social norms (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Reduce stigma and normalize retesting by explaining that it is a common practice for people to be aware of their HIV status and get tested often when they are at risk
  * I.e., don't be part of the small proportion that isn't getting regularly tested
  * Leverages social pressure to participate in retesting
  * Uses a relatable community member to deliver the message
  Interventions: Behavioral: Social norms messaging
- Empowerment/goal-setting (Experimental): A "nudge" message, based in behavioral economics theory, that adheres to the following core concepts:
  * Encouraging motivation of participants to set a goal for follow-up testing
  * Empowering individuals through promotion of HIV retesting
  Interventions: Behavioral: Empowerment messaging

INTERVENTIONS:
Behavioral: Risk assessment messaging — Participants who are randomized to the "HIV risk assessment" arm will receive a brief video message at their baseline visit, containing information related to HIV risk assessment core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the HIV risk assessment content category.
  Arms: HIV Risk Assessment
Behavioral: U=U messaging — Participants who are randomized to the "U=U" arm will receive a brief video message at their baseline visit, containing information related to U=U core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the U=U content category.
  Arms: U=U messaging
Behavioral: Healthy Living messaging — Participants who are randomized to the "Healthy Living" arm will receive a brief video message at their baseline visit, containing information related to Healthy Living core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Healthy Living content category.
  Arms: Healthy Living
Behavioral: Community benefits messaging — Participants who are randomized to the "Community benefits" arm will receive a brief video message at their baseline visit, containing information related to Community Benefits core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Community Benefits content category.
  Arms: Community benefits
Behavioral: Fresh start effect — Participants who are randomized to the "Fresh start effect" arm will receive a brief video message at their baseline visit, containing information related to Fresh Start core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Fresh start effect content category.
  Arms: Fresh start effect
Behavioral: Education-based messaging (#1) — Participants who are randomized to the "Education-based #1" arm will receive a brief video message at their baseline visit, containing information related to HIV education core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Education-based #1 content category.
  Arms: Education-based #1
Behavioral: Education-based #2 messaging (gamification) — Participants who are randomized to the "Education-based #2" arm will receive a brief video message at their baseline visit, containing information related to HIV education/gamification core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Education-based/gamification content category.
  Arms: Education-based #2
Behavioral: Default appointment messaging — Participants who are randomized to the "Default appointment" arm will receive a brief video message at their baseline visit, containing information related to Default Appointment core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Default Appointment content category.
  Arms: Default appointment
Behavioral: Reserved for you messaging — Participants who are randomized to the "Reserved for you" arm will receive a brief video message at their baseline visit, containing information related to the Reserved for you core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Reserved for you content category.
  Arms: Reserved for you
Behavioral: Social norms messaging — Participants who are randomized to the "Social norms" arm will receive a brief video message at their baseline visit, containing information related to Social Norms core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Social Norms content category.
  Arms: Social norms
Behavioral: Empowerment messaging — Participants who are randomized to the "Empowerment/goal setting" arm will receive a brief video message at their baseline visit, containing information related to Empowerment core concepts and encouraging them to return for a repeat HIV test. They will also receive brief SMS follow-up messages at 8 and 11 week after baseline reminding them about HIV retesting and re-emphasizing concepts from the Empowerment content category.
  Arms: Empowerment/goal-setting

SUMMARY:
In this pilot study, the investigators will determine the feasibility and acceptability of multiple low-cost behavioral interventions, designed with end-user input, to promote HIV retesting among adults in rural Kenya and Uganda who have higher risk of HIV exposure.

DETAILED DESCRIPTION:
HIV re-testing is crucial in ensuring early identification of disease to promote well-being of an individual as well as preventing onward spread of infection by treating those identified to have disease promptly. The proposed study aims to identify approaches that would encourage individuals aged 15 years and above at high risk of HIV infection to retest. This IBIS Megastudy pilot trial will pilot 11 intervention prototypes for acceptability, feedback, and implementation outcomes prior to using the interventions in a larger-scale Megastudy trial (main trial to be submitted as a separate CT.gov record).

ELIGIBILITY:
Inclusion Criteria:

* at least 15 years of age
* At increased risk of HIV infection (defined by self-reported risk [at least one of the following over the 3 months prior to enrollment: >1 sexual partner, known HIV-positive sexual partner, diagnosed with a sexually transmitted infection, or paid or received gifts or money in exchange for sex] or by Kenya or Uganda MoH criteria for priority group)
* Documented negative HIV antibody test within 7 days of enrollment
* No intent to migrate out of community in next 3 months
* Daily access to a mobile phone (required since some of the interventions will be delivered by phone)

Exclusion Criteria:

* HIV-positive

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
8-11 locally adapted nudge interventions for inclusion in an upcoming randomized-controlled trial (IBIS Megastudy RCT) | 9 months
  The primary outcome from this pilot trial will be 8-11 locally adapted nudge interventions, which will later be used in an upcoming RCT (IBIS Megastudy RCT) with a separate clinicaltrials.gov registration record (not yet entered). The final nudge interventions which will be developed through this pilot trial will include local language and content refinement of the video and SMS scripts.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Chamie, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (2):
- Kenya Medical Research Institution (KEMRI), Mbita, Kenya
- Infectious Diseases Research Collaboration (IDRC), Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share de-identified IPD from our baseline questionnaire, which includes questions about subject demographics and HIV risk.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 36 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP).